CLINICAL TRIAL: NCT02282397
Title: Multiple Daily Injections and Continuous Glucose Monitoring in Diabetes
Acronym: DIaMonD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DexCom, Inc. (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PTL-901148
Record Dates: First submitted 2014-10-29; First posted 2014-11-04 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1: SMBG (No Intervention): Type 1 or Type 2 diabetes mellitus subjects using SMBG testing and usual care for diabetes management. No intervention to be administered
- Phase 1: CGM (Other): Type 1 or Type 2 diabetes mellitus subjects using RT-CGM and SMBG testing for diabetes management. RT-CGM (Continuous Glucose Monitoring) is the intervention.
  Interventions: Device: Continuous Glucose Monitor
- Phase 2: CGM/MDI (No Intervention): Type 1 Diabetes Mellitus subjects using RT-CGM and injections for diabetes management.
- Phase 2: CGM/CSII (No Intervention): Type 1 Diabetes Mellitus subjects using RT-CGM and CSII for diabetes management.

INTERVENTIONS:
Device: Continuous Glucose Monitor — RT-CGM are adjunctive devices with glucose trend graphs and user-configurable low and high glucose alerts.
  Other Names: CGM; RT-CGM
  Arms: Phase 1: CGM

SUMMARY:
Evaluate if addition and use of real time continuous glucose monitoring (RT-CGM) improves glycemic outcome of patients using multiple daily injections (MDI) and self monitoring blood glucose (SMBG) testing, who are not at target glycemic control.

DETAILED DESCRIPTION:
The study design includes two cohorts that will be treated separately. Phase 1 will include two diabetes cohorts (Type 1 diabetes mellitus and Type 2 diabetes mellitus) who will be randomized independently into two groups, Group 1-CGM and Group 2-SMBG.

The Group-1 CGM cohort who have Type 1 diabetes mellitus will be eligible for Phase 2. Phase 2 will include a separate independent randomization of either MDI therapy (Group 1a- CGM/MDI) or CSII therapy (Group 1b-CGM/CSII).

Additional assessments will be made to evaluate the incremental benefits of changing the insulin delivery method from MDI to CSII in patients already using CGM.

Cost effectiveness and quality of life will be measured between the two groups in each phase.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 years or older
* Diagnosis of Type 1 diabetes mellitus or insulin-requiring Type 2 diabetes mellitus
* Followed regularly by a physician or diabetes educator
* Using multiple daily injections
* stable control of diabetes
* willing to wear a device such as pump or continuous glucose monitor

Exclusion Criteria:

* recent or planned use of non-insulin injectable hypoglycemic agents
* Pregnancy or planning to become pregnant during the study
* Medical conditions that make it inappropriate or unsafe to target an A1C of <7%
* Renal disease with Glomerular Filtration Rate <45
* Extensive skin changes/disease that precludes wearing the sensor on normal skin
* Known allergy to medical-grade adhesives
* Recent hospitalization or emergency room visit in the 6 months prior to screening resulting in primary diagnosis of uncontrolled diabetes

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2014-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Phase 1 (T1DM) - A1C | 6 months
  Change in A1C from baseline to 24 weeks
Phase 1 (T2DM) - A1C | 6 months
  Change in A1C from baseline to 24 weeks
Phase 2 (T1DM) | 6 months
  Change in % time in range 70-180 mg/dL from Phase 2 baseline to Phase 2 28 weeks

SECONDARY OUTCOMES:
Phase 1 (T1DM) - A1C Outcomes | 6 months
  % of subjects with A1C less than 7%
Phase 1 (T1DM) - A1C Outcomes | 6 months
  % of subjects with A1C less than 7.5%
Phase 1 (T1DM) - A1C Outcomes | 6 months
  % of subjects with a relative reduction in A1C greater than or equal to 10%
Phase 1 (T1DM) - A1C Outcomes | 6 months
  % of subjects with a reduction in A1C greater than or equal to 1%
Phase 1 (T1DM) - A1C Outcomes | 6 months
  % of subjects with a reduction in A1C greater than or equal to 1% or A1C less than 7%
Phase 1 (T1DM) - CGM Outcomes | 6 months
  Mean glucose (overall, daytime, and nighttime separately)
Phase 1 (T1DM) - CGM Outcomes | 6 months
  Glucose variability (overall, daytime, and nighttime separately)
Phase 1 (T1DM) - CGM Outcomes | 6 months
  % time in range 70-180 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T1DM) - CGM Outcomes | 6 months
  % time less than 70 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T1DM) - CGM Outcomes | 6 months
  % time less than 60 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T1DM) - CGM Outcomes | 6 months
  % time less than 50 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T1DM) - CGM Outcomes | 6 months
  % time greater than 180 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T1DM) - CGM Outcomes | 6 months
  % time greater than 250 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T1DM) - CGM Outcomes | 6 months
  % time greater than 300 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T1DM) - Hypoglycemia Awareness | 6 months
  Change in Clarke Hypoglycemia Unawareness score from baseline to 24 weeks
Phase 1 (T1DM) - SMBG Outcome | 6 months
  Change in SMBG frequency from baseline to 24 weeks
Phase 1 (T1DM) - QoL Outcomes | 6 months
  Quality of life changes from baseline to 24 weeks
Phase 1 (T1DM) - Cost Effectiveness | 6 months
  Cost effectiveness measured by the incremental cost-effectiveness ratio (ICER)
Phase 1 (T1DM) - Adverse Events | 6 months
  Change in the number of SH events from baseline to 24 weeks
Phase 1 (T1DM) - Adverse Events | 6 months
  Change in the number of DKA events from baseline to 24 weeks
Phase 1 (T1DM) - Body Weight | 6 months
  Change in body weight from baseline to 24 weeks
Phase 1 (T1DM) - Insulin Use Outcomes | 6 months
  Change in total daily insulin from baseline to 24 weeks
Phase 1 (T1DM) - Insulin Use Outcomes | 6 months
  Basal to bolus insulin ratio
Phase 1 (T1DM) - Insulin Use Outcomes | 6 months
  Change in the number of boluses/day from baseline to 24 weeks
Phase 1 (T2DM) - A1C Outcomes | 6 months
  % of subjects with A1C less than 7%
Phase 1 (T2DM) - A1C Outcomes | 6 months
  % of subjects with A1C less than 7.5%
Phase 1 (T2DM) - A1C Outcomes | 6 months
  % of subjects with a relative reduction in A1C greater than or equal to 10%
Phase 1 (T2DM) - A1C Outcomes | 6 months
  % of subjects with a reduction in A1C greater than or equal to 1% or A1C less than 7%
Phase 1 (T2DM) - A1C Outcomes | 6 months
  % of subjects with a reduction in A1C greater than or equal to 1%
Phase 1 (T2DM) - CGM Outcomes | 6 months
  Mean glucose (overall, daytime, and nighttime separately)
Phase 1 (T2DM) - CGM Outcomes | 6 months
  Glucose variability (overall, daytime, and nighttime separately)
Phase 1 (T2DM) - CGM Outcomes | 6 months
  % time in range 70-180 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T2DM) - CGM Outcomes | 6 months
  % time less than 70 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T2DM) - CGM Outcomes | 6 months
  % time less than 60 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T2DM) - CGM Outcomes | 6 months
  % time less than 50 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T2DM) - CGM Outcomes | 6 months
  % time greater than 180 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T2DM) - CGM Outcomes | 6 months
  % time greater than 250 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T2DM) - CGM Outcomes | 6 months
  % time greater than 300 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T2DM) - CGM Outcomes | 6 months
  Area above curve 70 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T2DM) - CGM Outcomes | 6 months
  Area under curve 180 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T2DM) - Hypoglycemia Awareness | 6 months
  Change in Clarke Hypoglycemia Unawareness score from baseline to 24 weeks
Phase 1 (T2DM) - SMBG | 6 months
  Change in SMBG frequency from baseline to 24 weeks
Phase 1 (T2DM) - QoL Outcomes | 6 months
  Quality of life changes from baseline to 24 weeks
Phase 1 (T2DM) - Cost Effectiveness | 6 months
  Cost effectiveness measured by the incremental cost-effectiveness ratio (ICER)
Phase 1 (T2DM) - Adverse Events | 6 months
  Change in the number of SH Events from baseline to 24 weeks
Phase 1 (T2DM) - Adverse Events | 6 months
  Change in the number of DKA Events from baseline to 24 weeks
Phase 1 (T2DM) - Body Weight | 6 months
  Change in body weight from baseline to 24 weeks
Phase 1 (T2DM) - Insulin Use Outcomes | 6 months
  Change in total daily insulin from baseline to 24 weeks
Phase 1 (T2DM) - Insulin Use Outcomes | 6 months
  Basal to bolus insulin ratio
Phase 1 (T2DM) - Insulin Use Outcomes | 6 months
  Change in the number of boluses/day from baseline to 24 weeks
Phase 2 (T1DM) - A1C Outcomes | 6 months
  Change in A1C from Phase 2 baseline to Phase 2 28 weeks
Phase 2 (T1DM) - A1C Outcomes | 6 months
  % of subjects with A1C less than 7%
Phase 2 (T1DM) - A1C Outcomes | 6 months
  % of subjects with A1C less than 7.5%
Phase 2 (T1DM) - A1C Outcomes | 6 months
  % of subjects with a relative reduction in A1C greater than or equal to 10%
Phase 2 (T1DM) - A1C Outcomes | 6 months
  % of subjects with a reduction in A1C greater than or equal to 1%
Phase 2 (T1DM) - A1C Outcomes | 6 months
  % of subjects with a reduction in A1C greater than or equal to 1% or A1C less than 7%
Phase 2 (T1DM) - CGM Outcomes | 6 months
  Mean glucose (overall, daytime, and nighttime separately)
Phase 2 (T1DM) - CGM Outcomes | 6 months
  Glucose variability (overall, daytime, and nighttime separately)
Phase 2 (T1DM) - CGM Outcomes | 6 months
  % time less than 70 mg/dL (overall, daytime, and nighttime separately)
Phase 2 (T1DM) - CGM Outcomes | 6 months
  % time less than 60 mg/dL (overall, daytime, and nighttime separately)
Phase 2 (T1DM) - CGM Outcomes | 6 months
  % time less than 50 mg/dL (overall, daytime, and nighttime separately)
Phase 2 (T1DM) - CGM Outcomes | 6 months
  % time greater than 180 mg/dL (overall, daytime, and nighttime separately)
Phase 2 (T1DM) - CGM Outcomes | 6 months
  % time greater than 250 mg/dL (overall, daytime, and nighttime separately)
Phase 2 (T1DM) - CGM Outcomes | 6 months
  % time greater than 300 mg/dL (overall, daytime, and nighttime separately)
Phase 2 (T1DM) - CGM Outcomes | 6 months
  Area above curve 70 mg/dL (overall, daytime, and nighttime separately)
Phase 2 (T1DM) - CGM Outcomes | 6 months
  Area above curve 180 mg/dL (overall, daytime, and nighttime separately)
Phase 2 (T1DM) - Hypoglycemia Awareness | 6 months
  Change in Clarke Hypoglycemia Unawareness score from Phase 2 baseline to Phase 2 28 weeks
Phase 2 (T1DM) - CGM Use | 6 months
  Change in frequency of CGM use from Phase 2 baseline to Phase 2 28 weeks
Phase 2 (T1DM) - SMBG | 6 months
  Change in SMBG frequency from Phase 2 baseline to Phase 2 28 weeks
Phase 2 (T1DM) - QoL Outcomes | 6 months
  Quality of life changes from Phase 2 baseline to Phase 2 28 weeks
Phase 2 (T1DM) - Cost Effectiveness | 6 months
  Cost effectiveness measured by the incremental cost-effectiveness ratio (ICER)
Phase 2 (T1DM) - Adverse Events | 6 months
  Change in the number of SH Events from Phase 2 baseline to Phase 2 28 weeks
Phase 2 (T1DM) - Adverse Events | 6 months
  Change in the number of DKA Events from Phase 2 baseline to Phase 2 28 weeks
Phase 2 (T1DM) - Body Weight | 6 months
  Change in body weight from Phase 2 baseline to Phase 2 28 weeks
Phase 2 (T1DM) - Insulin Use Outcomes | 6 months
  Change in total daily insulin from Phase 2 baseline to Phase 2 28 weeks
Phase 2 (T1DM) - Insulin Use Outcomes | 6 months
  Basal to bolus insulin ratio
Phase 2 (T1DM) - Insulin Use Outcomes | 6 months
  Change in the number of boluses/day from Phase 2 baseline to Phase 2 28 weeks

OTHER OUTCOMES:
Phase 1 (T1DM) - Post-Hoc CGM Outcomes | 6 months
  Area above curve 70 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T1DM) - Post-Hoc CGM Outcomes | 6 months
  Area under curve 180 mg/dL (overall, daytime, and nighttime separately)
Phase 1 (T2DM) - Post-Hoc A1C Outcome | 6 months
  % of subjects with a reduction in A1C greater than or equal to 0.5%

CONTACTS AND LOCATIONS:
Overall Officials: David Price, MD, Study Director — DexCom, Inc.
Locations (29):
- United States (26):
  - Marin Endocrine Care & Research, Greenbrae, California
  - Coastal Metabolic Research Centre, Ventura, California
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Laureate Medical Group at Northside, LLC, Atlanta, Georgia
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Physicians Research Associates, LLC, Lawrenceville, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Rocky Mountain Diabetes & Osteoporosis Center, Idaho Falls, Idaho
  - Iowa Diabetes & Endocrinology Research Center, Des Moines, Iowa
  - Joslin Diabetes Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Diabetes & Endocrine Associates, PC, Omaha, Nebraska
  - Accent Clinical Research, Las Vegas, Nevada
  - Albany Medical College, Albany, New York
  - Mountain Diabetes and Endocrine Center, Asheville, North Carolina
  - Legacy Research Institute, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Amarillo Medical Specialists, LLP, Amarillo, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Diabetes and Glandular Disease, San Antonio, Texas
  - Consano Clinical Research, San Antonio, Texas
  - Advanced Research Associates, Ogden, Utah
  - Granger Medical Clinic, Riverton, Utah
- Canada (3):
  - LMC Clinical Research, Barrie, Ontario
  - LMC Clinical Research, Thornhill, Ontario
  - LMC Clinical Research, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hermanns N, Ehrmann D, Heinemann L, Freckmann G, Waldenmaier D, Calhoun P. Real-Time Continuous Glucose Monitoring Can Predict Severe Hypoglycemia in People with Type 1 Diabetes: Combined Analysis of the HypoDE and DIAMOND Trials. Diabetes Technol Ther. 2022 Sep;24(9):603-610. doi: 10.1089/dia.2022.0130. Epub 2022 Jun 10. PMID 35604794
- [Derived] Puhr S, Welsh JB, Bauza CE, Walker TC. Patients with Type 2 Diabetes and Residual Insulin Secretory Capacity Realize Glycemic Benefits from Real-Time Continuous Glucose Monitoring. J Diabetes Sci Technol. 2021 Jul;15(4):965-967. doi: 10.1177/19322968211007880. Epub 2021 Apr 15. No abstract available. PMID 33855888
- [Derived] Calhoun P, Price D, Beck RW. Glycemic Improvement Using Continuous Glucose Monitoring by Baseline Time in Range: Subgroup Analyses from the DIAMOND Type 1 Diabetes Study. Diabetes Technol Ther. 2021 Mar;23(3):230-233. doi: 10.1089/dia.2020.0471. Epub 2020 Oct 20. PMID 33006904
- [Derived] Puhr S, Calhoun P, Welsh JB, Walker TC. The Effect of Reduced Self-Monitored Blood Glucose Testing After Adoption of Continuous Glucose Monitoring on Hemoglobin A1c and Time in Range. Diabetes Technol Ther. 2018 Aug;20(8):557-560. doi: 10.1089/dia.2018.0134. Epub 2018 Jul 23. PMID 30036082
- [Derived] Beck RW, Riddlesworth TD, Ruedy K, Ahmann A, Haller S, Kruger D, McGill JB, Polonsky W, Price D, Aronoff S, Aronson R, Toschi E, Kollman C, Bergenstal R; DIAMOND Study Group. Continuous Glucose Monitoring Versus Usual Care in Patients With Type 2 Diabetes Receiving Multiple Daily Insulin Injections: A Randomized Trial. Ann Intern Med. 2017 Sep 19;167(6):365-374. doi: 10.7326/M16-2855. Epub 2017 Aug 22. PMID 28828487
- [Derived] Beck RW, Riddlesworth TD, Ruedy KJ, Kollman C, Ahmann AJ, Bergenstal RM, Bhargava A, Bode BW, Haller S, Kruger DF, McGill JB, Polonsky W, Price D, Toschi E; DIAMOND Study Group. Effect of initiating use of an insulin pump in adults with type 1 diabetes using multiple daily insulin injections and continuous glucose monitoring (DIAMOND): a multicentre, randomised controlled trial. Lancet Diabetes Endocrinol. 2017 Sep;5(9):700-708. doi: 10.1016/S2213-8587(17)30217-6. Epub 2017 Jul 12. PMID 28711468
- [Derived] Riddlesworth T, Price D, Cohen N, Beck RW. Hypoglycemic Event Frequency and the Effect of Continuous Glucose Monitoring in Adults with Type 1 Diabetes Using Multiple Daily Insulin Injections. Diabetes Ther. 2017 Aug;8(4):947-951. doi: 10.1007/s13300-017-0281-4. Epub 2017 Jun 14. PMID 28616804
- [Derived] Polonsky WH, Hessler D, Ruedy KJ, Beck RW; DIAMOND Study Group. The Impact of Continuous Glucose Monitoring on Markers of Quality of Life in Adults With Type 1 Diabetes: Further Findings From the DIAMOND Randomized Clinical Trial. Diabetes Care. 2017 Jun;40(6):736-741. doi: 10.2337/dc17-0133. Epub 2017 Apr 7. PMID 28389582
- [Derived] Beck RW, Riddlesworth T, Ruedy K, Ahmann A, Bergenstal R, Haller S, Kollman C, Kruger D, McGill JB, Polonsky W, Toschi E, Wolpert H, Price D; DIAMOND Study Group. Effect of Continuous Glucose Monitoring on Glycemic Control in Adults With Type 1 Diabetes Using Insulin Injections: The DIAMOND Randomized Clinical Trial. JAMA. 2017 Jan 24;317(4):371-378. doi: 10.1001/jama.2016.19975. PMID 28118453